CLINICAL TRIAL: NCT00557869
Title: Optimization of Native Cardiac-MR Protocols
Brief Title: Optimization of Cardiac-MR Protocols
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Ursula Reiter, PhD, Medical University of Graz
Other Study IDs: CMR-02-TECH-01
Record Dates: First submitted 2007-11-13; First posted 2007-11-14 (Estimated); Last update posted 2011-12-20 (Estimated); Status verified 2011-12

CONDITIONS: Sequence Optimization; Protocol Optimization; Normal Values; Feasibility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of the present study is the optimization of various magnetic resonance (MR) investigation protocols of the heart and the lung without contrast agent application as well as the generation of normal values from cardiac MR images. One of the main problems in cardiac MR investigations is the strong dependence of the achieved image quality on optimal settings of sequence parameters and anatomical and physiological situations with special emphasis on phase-contrast imaging and other cine-techniques.

DETAILED DESCRIPTION:
Time optimized and well organized MR protocols for the cardiac and lung investigations are evaluated on normal subjects with special respect to following topics:

1. Localization: Definition of standardized anatomic imaging planes with special respect to the right ventricle.
2. Morphological imaging: Optimization of spin-echo and gradient-echo sequences for various heart frequencies and breath-hold abilities. Investigation of the effect of various preparation pulses. Optimization of the signal-to-noise ratio for morphological cardiac imaging. Evaluation and optimization of various breathing and breath-hold (with and without navigator) ECG and pulse triggered sequences.
3. Cardiac and lung function: Optimization of gradient-echo sequences for various heart frequencies and breath-hold abilities. Evaluation of pulse-triggered function analysis and optimization of free breathing protocols. Optimization of tagging techniques. Evaluation of the pulsatile flow in lung vessels. Acquisition of age depended normal data of cardiac and lung function.
4. Coronary imaging: Definition of standardized anatomic imaging planes to monitor coronary arteries (single oblique, volume targeted). Optimization of acquisition window with respect to various heart frequencies. Evaluation of the influence of the position of the navigator and tracking factor on image quality. Optimization of a pulse triggered protocol. Evaluation of black-blood coronary imaging and visualization of the lumen and wall of coronary arteries.
5. Phase contrast techniques: Optimization of imaging planes, time resolution and spatial resolution of flow measurements in the heart, in the vessels around the heart, lung vessels and coronary arteries. Evaluation of retrospective and prospective gating with respect to the heart frequency. Evaluation of normal values in 1-dimensional, 2-dimensional and 3-dimensional time resolved flow measurements.
6. Single-Shot Imaging: Evaluation of signal intensity and stability of single shot techniques with and without preparation pulses. Optimization of real-time image acquisition.
7. Parallel acquisition and breath-hold time optimization: Evaluation of impact of echo-sharing and parallel acquisition on image quality. Optimization of short-breath-hold protocols.

ELIGIBILITY:
Inclusion Criteria:

* No history of cardiac or pulmonary diseases

Exclusion Criteria:

* MRI exclusion criteria

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2002-10; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gert Reiter, DI Dr., Principal Investigator — Siemens Medical Solutions; Ursula Reiter, DI Dr., Principal Investigator — University Hospital Graz
Locations (1):
- Medical Unitersity Graz, Allgemeine Radiologische Diagnostik, Graz, Stmk, Austria

REFERENCES:
- [Result] Reiter G, Reiter U, Bergmann P, Rienmuller R. MR imaging-based port placement planning for totally endoscopic coronary artery bypass grafting. Interact Cardiovasc Thorac Surg. 2004 Jun;3(2):341-5. doi: 10.1016/j.icvts.2004.01.015. PMID 17670255
- [Result] Reiter G, Reiter U, Rienmuller R, Gagarina N, Ryabikin A. On the value of geometry-based models for left ventricular volumetry in magnetic resonance imaging and electron beam tomography: a Bland-Altman analysis. Eur J Radiol. 2004 Nov;52(2):110-8. doi: 10.1016/j.ejrad.2003.10.003. PMID 15489068
- [Result] Reiter G, Reiter U, Kovacs G, Kainz B, Schmidt K, Maier R, Olschewski H, Rienmueller R. Magnetic resonance-derived 3-dimensional blood flow patterns in the main pulmonary artery as a marker of pulmonary hypertension and a measure of elevated mean pulmonary arterial pressure. Circ Cardiovasc Imaging. 2008 Jul;1(1):23-30. doi: 10.1161/CIRCIMAGING.108.780247. PMID 19808511